CLINICAL TRIAL: NCT07042984
Title: RET-US Cohort: Prospective Evaluation of an AI-Ultrasound Model for Detecting RET Gene Alterations and Predicting Lateral Cervical Lymph-Node Metastasis in Papillary Thyroid Carcinoma
Brief Title: RET-US Study - Ultrasound-Based Prediction of RET Alterations and Lateral-Neck Metastasis in Thyroid Cancer
Acronym: RET-US
Status: Not yet recruiting | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Bo Wang,MD, Director & Head of Thyroid Surgery, Principal Investigator, Clinical Professor, Fujian Medical University Union Hospital
Other Study IDs: RET-US
Record Dates: First submitted 2025-06-21; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Papillary Thyroid Carcinoma; Thyroid Neoplasms; RET Proto-Oncogene Mutation; Lymphatic Metastasis
Keywords: Ultrasound Radiomics; Artificial Intelligence; RET Fusion; BRAF V600E; Lateral Neck Metastasis; Deep Learning Model; 11-Gene Panel
MeSH Terms: conditions — Thyroid Cancer, Papillary; Thyroid Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — FNA cytology and paraffin blocks are stored and include DNA extraction for the 11-gene panel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Thyroid Cancer Cohort: Consecutive adults (18-75 y) with ultrasound-suspected papillary thyroid carcinoma scheduled for surgery. Each participant undergoes standard pre-operative ultrasound, rapid 14-gene next-generation sequencing (NGS) panel, and blinded AI analysis of the ultrasound images. No treatment allocation is made; data are collected prospectively to validate the AI model's ability to detect RET alterations and predict lateral-neck lymph-node metastasis.
  Interventions: Diagnostic Test: AI-Ultrasound RET Prediction

INTERVENTIONS:
Diagnostic Test: AI-Ultrasound RET Prediction — Deep-learning algorithm that analyses thyroid ultrasound DICOM images and outputs a probability score for RET gene alteration and lateral-neck lymph-node metastasis; run offline, results blinded to treating surgeons.

SUMMARY:
Why is this study being done? RET gene alterations occur in only 5-10 % of papillary thyroid cancers, but they can change how surgeons treat the disease. Gene testing is costly and not always performed, so many RET-positive tumours are missed. Researchers have built a computer program (artificial-intelligence or "AI" model) that reads routine thyroid ultrasound images and predicts whether the tumour carries a RET alteration and whether the cancer has already spread to lymph-nodes in the side of the neck.

What will happen in this study?

About 800 adults who are scheduled for thyroid-cancer surgery will take part. Each participant will:

* have a standard pre-operative ultrasound exam (no extra scanning time),
* give a routine fine-needle sample for a 14-gene panel test (results in 24 h), and
* allow the AI model to analyse the ultrasound images in the background. Doctors making treatment decisions will not see the AI result. After surgery, the research team will compare the AI predictions with the gene-panel result and the final pathology report.

Main goal: To find out how accurately the AI model detects RET alterations. Secondary goals: To measure the model's ability to predict lymph-node spread, and to compare costs between ultrasound-only prediction and full gene testing.

Benefits and risks: Participants will receive the current standard of care; there is no added risk beyond the usual ultrasound and needle biopsy. The study could lead to faster, less expensive ways to identify high-risk thyroid cancers in the future.

DETAILED DESCRIPTION:
Background RET rearrangements or point mutations drive a minority of papillary thyroid carcinomas (PTC) yet are associated with aggressive behaviour and may qualify patients for selective RET inhibitors. Because of low prevalence, RET testing is often omitted, resulting in under-recognition. Recent work shows that high-resolution ultrasound contains radiomic signatures linked to tumour genotypes. A deep-learning model (EfficientNet-B3 backbone with dual segmentation + multi-label heads) was trained on 1 000 retrospectively collected cases, including 74 RET-positive tumours augmented with GAN-based synthetic images, achieving an AUC of 0.87 for RET prediction in internal cross-validation.

Objectives Primary: validate the AI model's area under the receiver-operating characteristic curve (AUC) for RET alteration detection in a prospective cohort.

Secondary: (i) sensitivity/specificity for RET; (ii) accuracy for predicting lateral-neck (pN1b) metastasis; (iii) incremental cost per correct RET diagnosis; (iv) concordance between AI probability score and lymph-node burden.

Design Single-arm, prospective observational cohort (n = 800). Consecutive eligible patients will undergo: (1) routine pre-operative thyroid ultrasound; (2) upload of DICOM files to a cloud inference server; (3) rapid 14-gene next-generation sequencing panel on FNA or paraffin tissue (includes RET fusions KIF5B, CCDC6, NCOA4 and point mutations M918T, V804). Surgeons remain blinded to AI output. Surgical specimens provide ground truth for pN staging. Data captured in REDCap; statistical analysis uses DeLong test for AUC and McNemar test for paired accuracy.

Eligibility Adults 18-75 y with radiologically suspected PTC, planned thyroidectomy, and consent for gene testing. Exclusions: re-operative neck, medullary/anaplastic carcinoma, pregnancy, eGFR < 30 mL min-¹ 1.73 m-².

Sample Size With expected RET prevalence 6 % and target AUC ≥ 0.80 vs null 0.50, 800 cases provide 90 % power (α = 0.05).

Ethics & Oversight IRB approved; minimal-risk diagnostic study. Ultrasound and FNA are standard-of-care; AI inference uses de-identified images. Results will be disseminated via peer-reviewed journals and conference presentations.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, able to provide written informed consent.
* Pre-operative ultrasound findings highly suggestive of papillary thyroid carcinoma.
* Planned thyroidectomy (any extent) at a participating institution.
* Willing to undergo rapid 11-gene next-generation sequencing (NGS) panel and allow use of ultrasound DICOM images for AI analysis.

Exclusion Criteria:

* Prior thyroid or major neck surgery.
* Known medullary thyroid carcinoma, anaplastic carcinoma, or metastatic disease outside the neck.
* Multiple endocrine neoplasia (MEN) syndromes or clinical suspicion of multi-gland disease.
* Pregnant or breastfeeding.
* Severe renal impairment (eGFR < 30 mL/min/1.73 m²) or other condition that precludes surgery or gene testing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adults with ultrasound-suspected papillary thyroid carcinoma scheduled for thyroidectomy at participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Area Under the ROC Curve (AUC) for AI-Ultrasound Detection of RET Alterations | Date of surgery (assessment completed when gene-panel result is available)
  The receiver-operating-characteristic area under the curve comparing the AI-generated probability score against the reference 14-gene next-generation sequencing (NGS) result for RET fusion or point mutation. AUC calculated with 95 % confidence interval via DeLong method.

SECONDARY OUTCOMES:
Sensitivity and Specificity of AI-Ultrasound for Detecting RET Alterations | Date of surgery (assessment completed when NGS result is available)
  Using the threshold that maximized the Youden index in the development set, calculate sensitivity (true-positive rate) and specificity (true-negative rate) of the AI model versus 11-gene NGS reference for RET fusion or point mutation. Results reported with 95 % confidence intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, FJ, China

IPD SHARING:
Plan to Share IPD: Undecided